CLINICAL TRIAL: NCT04777175
Title: A Retrospective Study: Evaluation of the Efficacy of Immunotherapy With Rare Mutations in Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Yongchang Zhang (Other)
Collaborators: Hunan Province Tumor Hospital (Other)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Other Study IDs: IRMLC
Record Dates: First submitted 2021-02-27; First posted 2021-03-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunization, Passive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- KRAS mutation: patients carry with KRAS mutation
  Interventions: Drug: immunity therapy
- ALK fusion: patients carry with ALK fusion
  Interventions: Drug: immunity therapy
- ERBB2 mutation: patients carry with ERBB2 mutation
  Interventions: Drug: immunity therapy
- MET skipping/amplication: patients carry with MET skipping/amplication
  Interventions: Drug: immunity therapy
- RET fusion: patients carry with RET fusion
  Interventions: Drug: immunity therapy
- BRAF mutation: patients carry with BRAF mutation
  Interventions: Drug: immunity therapy

INTERVENTIONS:
Drug: immunity therapy — The patient receives immunotherapy

SUMMARY:
In advanced non-small cell lung cancer, there will be some rare mutations, such as ALK, KRAS, etc. The efficacy of these immunotherapies on these different rare mutations has not been reported. Therefore, we conducted this retrospective clinical study to explore the efficacy of immunotherapy for different rare mutations.

ELIGIBILITY:
Inclusion Criteria:

* 1.Diagnosed as advanced non-small cell lung cancer
* 2.Confirmed as KARS, ALK, ERBB2, MET, RET, BRAF mutation

Exclusion Criteria:

* The patient is diagnosed with small cell lung cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-small-cell lung cancer carrying KRAS, ALK, ERBB2, MET, RET, BRAF mutation.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-12 (Estimated)

PRIMARY OUTCOMES:
PFS | January 2021- January 2021 (1 year)
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Hunan Cancer hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No